CLINICAL TRIAL: NCT00811954
Title: The ARDENT Study: Atazanavir, Raltegravir, or Darunavir With Emtricitabine/Tenofovir for Naive Treatment
Brief Title: Comparative Study of Three NNRTI-Sparing HAART Regimens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Bristol-Myers Squibb (Industry); Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry); Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5257; 1U01AI068636 (NIH)
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infection
Keywords: Treatment naive; Treatment inexperienced
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium; Darunavir; Ritonavir; Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: ATV/RTV + FTC/TDF (Experimental): Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF), ritonavir (RTV), and atazanavir (ATV) to be taken orally, once daily.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Ritonavir; Drug: Atazanavir
- Arm B: RAL + FTC/TDF (Experimental): FTC/TDF orally, once daily, and raltegravir (RAL) orally, twice daily.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Raltegravir
- Arm C: DRV/RTV + FTC/TDF (Experimental): FTC/TDF, darunavir (DRV), and RTV, orally, once daily.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Darunavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Emtricitabine/tenofovir disoproxil fumarate — 200 mg emtricitabine/300 mg tenofovir disoproxil fumarate taken orally daily. A combination drug of two nucleoside reverse transcriptase inhibitors (NRTIs).
  Other Names: TDF/FTC
Drug: Raltegravir — 400 mg taken orally twice daily. An integrase inhibitor (INI).
  Other Names: RAL
  Arms: Arm B: RAL + FTC/TDF
Drug: Darunavir — 800 mg taken orally once daily. A protease inhibitor (PI).
  Other Names: DRV
  Arms: Arm C: DRV/RTV + FTC/TDF
Drug: Ritonavir — 100 mg taken orally once daily. A protease inhibitor (PI).
  Other Names: RTV
  Arms: Arm A: ATV/RTV + FTC/TDF; Arm C: DRV/RTV + FTC/TDF
Drug: Atazanavir — 300 mg taken orally once daily. A protease inhibitor (PI).
  Other Names: ATV
  Arms: Arm A: ATV/RTV + FTC/TDF

SUMMARY:
The U.S. Department of Health and Human Services (HHS) guidelines recommend that HIV infected patients who have never received anti-HIV therapy be treated with a triple drug regimen. The most commonly prescribed and successful regimen contains the medication efavirenz (EFV). However, this regimen may not be an option for everyone, hence alternative regimens are needed.

This study was designed to look at how well different combinations of anti-HIV drugs work to decrease the amount of HIV in the blood (viral load) of and allow immune system recovery in people who have never received anti-HIV therapy. This study also examined drug tolerability and safety for the various drug combinations.

DETAILED DESCRIPTION:
Of the five anti-HIV drug classes, four were recommended as first-line regimens for patients who have never received anti-HIV treatment before (treatment naive): nucleoside reverse transcriptase inhibitors (NRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs), Integrase Inhibitors (INIs) and protease inhibitors (PIs). The U.S. Department of Health and Human Services (HHS) guidelines recommend that treatment-naive HIV infected patients be treated with a triple drug regimen that includes 2 NRTIs + 1 NNRTI, 2 NRTIs + INI, or 2 NRTIs + 1 PI as their initial treatment regimen.

According to data, an efavirenz (EFV)-containing regimen (2 NRTIs + 1 NNRTI, with EFVas the NNRTI) requires fewer pills for the patient, has mild and few side effects, and is more effective in reducing viral load than other regimens, making it the preferred choice for most patients. However, for some patients, an EFV-containing regimen is not feasible due to side effects, acquired NNRTI-resistant HIV virus, or other undesirable effects. For these patients, it is necessary to find alternative regimens with comparable safety and efficacy. This study examined how well different combinations of anti-HIV drugs work, including safety and drug tolerability for various combinations.

This was a phase III, prospective, randomized study. Participants was randomly assigned to one of three different groups (treatment arms)-A, B, or C -each representing a different drug combination regimen, none of which contained an NNRTI.

Arm A: Atazanavir (ATV) + Ritonavir (RTV) + Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF)

Arm B: Raltegravir (RAL) + FTC/TDF

Arm C: Darunavir (DRV) + RTV + FTC/TDF

The duration of this study was between 96 and 192 weeks, depending on when the participant enrolled. There were a total of 1,809 participants, approximately 600 per treatment arm. Screening and pre-entry evaluations must occur prior to the participant starting any study medication, treatments, or interventions. Participants were randomly assigned to their treatment groups at the entry visit and must begin treatment within 72 hours of randomization. Participants was told which group they were in and what medications they were administered. The study drugs were distributed at entry. All drugs were provided by the study with the exception of RTV, which would have to be obtained through the participant's primary care physician (Group A or C). If a participant was unable to tolerate any of the study medications during the course of the study then their doctor could switch them to another regimen.

During the study, participants was asked to return to the clinic at Weeks 4, 8, 16, 24, 36, and 48 and then every 16 weeks until the end of the study. They were also contacted by telephone during Week 2 to check on their status. Visits were last about 1 hour. At most visits, participants had a physical exam and answered questions about any medications they were taken. Additionally, participants completed questionnaires addressing their smoking and alcohol habits, had blood drawn, and were asked to give urine samples. At some visits, participants had to come to the clinic without having eaten for 8 hours. If the participant was female and able to become pregnant, a pregnancy test might be given at any visit if pregnancy was suspected.

Some participants of A5257 were asked to participate in an optional metabolic substudy A5260s. This substudy took place at only some study sites and continued last up to 144 weeks, including time on A5257. The primary focus of this substudy was to examine carotid artery intima-media thickness (CIMT) as it relates to both RTV- and RAL-containing regimens. Randomization, stratification, treatment assignments, and study visits were as per A5257.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* No evidence of any exclusionary mutations defined as any major NRTI or PI resistance-associated mutation on any genotype or evidence of significant NRTI or PI resistance on any phenotype performed at any time prior to study entry. NNRTI-associated resistance mutations are not excluded. More information on this criterion can be found in the study protocol.
* No prior anti-HIV therapy. More information on this criterion can be found in the study protocol.
* Viral load is 1000 copies/mL or higher, as measured within 90 days prior to study entry
* Certain laboratory values obtained within 60 days prior to study entry
* Ability to obtain RTV by prescription
* Completed cardiovascular risk assessment. More information on this criterion can be found in the study protocol.
* Must agree to use acceptable forms of contraception while receiving study drugs and for 6 weeks after stopping the medications. More information on this criterion is available in the protocol.
* Negative pregnancy test within 72 hours before initiating antiretroviral medication
* Participating in research at any AIDS Clinical Trial Group (ACTG) clinical research site or select International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) group sites
* Ability and willingness of subject or legal guardian/representative to give written informed consent

Exclusion Criteria:

* Use of immunomodulators, HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. Those using stable physiologic glucocorticoid doses, a short course of pharmacologic glucocorticoid, corticosteroids for acute therapy treating an opportunistic infection, inhaled or topical corticosteroids, or granulocyte-colony stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) will not be excluded.
* Known allergy or sensitivity to study drugs or their ingredients. A history of sulfa allergy is not excluded.
* Any condition that, in the opinion of the investigator, would compromise the participant's ability to participate in the study
* Serious illness requiring systemic treatment and/or hospitalization until participant either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 7 days prior to study entry
* Requirement for any current medications that are prohibited with any study drugs
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical illness
* Any prior use of entecavir for treatment of hepatitis B for greater than 8 weeks while the participant was known to be HIV infected
* Presence of decompensated cirrhosis
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1814 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Lennox, MD, Study Chair — Emory HIV/AIDS CTU; Judith Silverstein Currier, MD, MSc, Study Chair — UCLA AIDS Prevention & Treatment CTU; Raphael Landovitz, MD, MSc, Study Chair — UCLA AIDS Prevention & Treatment CTU; Igho Ofotokun, MD, Study Chair — Emory HIV/AIDS CTU
Locations (57):
- United States (55):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Miller Children's Hospital, Long Beach, California
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida Childrens Diagnostic & Treatment Cen (5055), Fort Lauderdale, Florida
  - University of Florida Jacksonville (5051), Jacksonville, Florida
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Tulane University New Orleans NICHD CRS (5095), New Orleans, Louisiana
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital CRS, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Wayne State Univ. CRS, Detroit, Michigan
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Washington U CRS, St Louis, Missouri
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - Cornell CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Metropolitan Hospital, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - AIDS Care CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS (5040), Stony Brook, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - Metro Health CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - The Research & Education Group- Portland CRS (31474), Portland, Oregon
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - Trinity Health and Wellness Center, Dallas, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS, Rio Piedras
  - Puerto Rico-AIDS CRS, San Juan

REFERENCES:
- [Background] Bartlett JA, Chen SS, Quinn JB. Comparative efficacy of nucleoside/nucleotide reverse transcriptase inhibitors in combination with efavirenz: results of a systematic overview. HIV Clin Trials. 2007 Jul-Aug;8(4):221-6. doi: 10.1310/hct0804-221. PMID 17720662
- [Background] Duvivier C, Ghosn J, Assoumou L, Soulie C, Peytavin G, Calvez V, Genin MA, Molina JM, Bouchaud O, Katlama C, Costagliola D; ANRS 121 study group. Initial therapy with nucleoside reverse transcriptase inhibitor-containing regimens is more effective than with regimens that spare them with no difference in short-term fat distribution: Hippocampe-ANRS 121 Trial. J Antimicrob Chemother. 2008 Oct;62(4):797-808. doi: 10.1093/jac/dkn278. Epub 2008 Jul 18. PMID 18641035
- [Background] Markowitz M, Nguyen BY, Gotuzzo E, Mendo F, Ratanasuwan W, Kovacs C, Prada G, Morales-Ramirez JO, Crumpacker CS, Isaacs RD, Gilde LR, Wan H, Miller MD, Wenning LA, Teppler H; Protocol 004 Part II Study Team. Rapid and durable antiretroviral effect of the HIV-1 Integrase inhibitor raltegravir as part of combination therapy in treatment-naive patients with HIV-1 infection: results of a 48-week controlled study. J Acquir Immune Defic Syndr. 2007 Oct 1;46(2):125-33. doi: 10.1097/QAI.0b013e318157131c. PMID 17721395
- [Background] Molina JM, Andrade-Villanueva J, Echevarria J, Chetchotisakd P, Corral J, David N, Moyle G, Mancini M, Percival L, Yang R, Thiry A, McGrath D; CASTLE Study Team. Once-daily atazanavir/ritonavir versus twice-daily lopinavir/ritonavir, each in combination with tenofovir and emtricitabine, for management of antiretroviral-naive HIV-1-infected patients: 48 week efficacy and safety results of the CASTLE study. Lancet. 2008 Aug 23;372(9639):646-55. doi: 10.1016/S0140-6736(08)61081-8. PMID 18722869
- [Derived] Hughey CM, Vuong BW, Ribaudo HB, Mitchell CCK, Korcarz CE, Hodis HN, Currier JS, Stein JH. Grayscale Ultrasound Texture Features of Carotid and Brachial Arteries in People With HIV Infection Before and After Antiretroviral Therapy. J Am Heart Assoc. 2022 Mar;11(5):e024142. doi: 10.1161/JAHA.121.024142. Epub 2022 Feb 18. PMID 35179037
- [Derived] Li B, Veturi Y, Verma A, Bradford Y, Daar ES, Gulick RM, Riddler SA, Robbins GK, Lennox JL, Haas DW, Ritchie MD. Tissue specificity-aware TWAS (TSA-TWAS) framework identifies novel associations with metabolic, immunologic, and virologic traits in HIV-positive adults. PLoS Genet. 2021 Apr 26;17(4):e1009464. doi: 10.1371/journal.pgen.1009464. eCollection 2021 Apr. PMID 33901188
- [Derived] Bares SH, Smeaton LM, Scott SE, Smith BA, Godfrey C, McComsey GA. The Association Between Weight Gain, Sex, and Immune Activation Following the Initiation of Antiretroviral Therapy. J Infect Dis. 2021 Nov 22;224(10):1765-1774. doi: 10.1093/infdis/jiab210. PMID 33870433
- [Derived] McComsey GA, Moser C, Currier J, Ribaudo HJ, Paczuski P, Dube MP, Kelesidis T, Rothenberg J, Stein JH, Brown TT. Body Composition Changes After Initiation of Raltegravir or Protease Inhibitors: ACTG A5260s. Clin Infect Dis. 2016 Apr 1;62(7):853-62. doi: 10.1093/cid/ciw017. Epub 2016 Jan 20. PMID 26797215
- [Derived] Kelesidis T, Tran TT, Stein JH, Brown TT, Moser C, Ribaudo HJ, Dube MP, Murphy R, Yang OO, Currier JS, McComsey GA. Changes in Inflammation and Immune Activation With Atazanavir-, Raltegravir-, Darunavir-Based Initial Antiviral Therapy: ACTG 5260s. Clin Infect Dis. 2015 Aug 15;61(4):651-60. doi: 10.1093/cid/civ327. Epub 2015 Apr 22. PMID 25904376
- [Derived] Ofotokun I, Na LH, Landovitz RJ, Ribaudo HJ, McComsey GA, Godfrey C, Aweeka F, Cohn SE, Sagar M, Kuritzkes DR, Brown TT, Patterson KB, Para MF, Leavitt RY, Villasis-Keever A, Baugh BP, Lennox JL, Currier JS; AIDS Clinical Trials Group (ACTG) A5257 Team. Comparison of the metabolic effects of ritonavir-boosted darunavir or atazanavir versus raltegravir, and the impact of ritonavir plasma exposure: ACTG 5257. Clin Infect Dis. 2015 Jun 15;60(12):1842-51. doi: 10.1093/cid/civ193. Epub 2015 Mar 12. PMID 25767256
- [Derived] Lennox JL, Landovitz RJ, Ribaudo HJ, Ofotokun I, Na LH, Godfrey C, Kuritzkes DR, Sagar M, Brown TT, Cohn SE, McComsey GA, Aweeka F, Fichtenbaum CJ, Presti RM, Koletar SL, Haas DW, Patterson KB, Benson CA, Baugh BP, Leavitt RY, Rooney JF, Seekins D, Currier JS; ACTG A5257 Team. Efficacy and tolerability of 3 nonnucleoside reverse transcriptase inhibitor-sparing antiretroviral regimens for treatment-naive volunteers infected with HIV-1: a randomized, controlled equivalence trial. Ann Intern Med. 2014 Oct 7;161(7):461-71. doi: 10.7326/M14-1084. PMID 25285539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at AIDS Clinical Trials Units in the United States and Puerto Rico. Recruitment occurred between May 22, 2009 (date first subject was randomized) and June 9, 2011 (date last subject was randomized).
Pre-assignment Details: 1814 were randomized 1:1:1 to treatment arms A, B, and C. Results reported for 1809 eligible participants; 5 were subsequently found ineligible and excluded from all analyses.
Groups:
- Arm A: ATV/RTV + FTC/TDF: Emtricitabine/tenofovir disoproxil fumarate (FTC/TDF), ritonavir (RTV), and atazanavir (ATV) to be taken orally, once daily.
  Emtricitabine/tenofovir disoproxil fumarate: A combination drug of two nucleoside reverse transcriptase inhibitors (NRTIs) Ritonavir: A protease inhibitor (PI) Atazanavir: A protease inhibitor (PI)
- Arm B: RAL + FTC/TDF: FTC/TDF orally, once daily, and raltegravir (RAL) orally, twice daily.
  Emtricitabine/tenofovir disoproxil fumarate: A combination drug of two nucleoside reverse transcriptase inhibitors (NRTIs) Raltegravir: An integrase inhibitor (INI)
- Arm C: DRV/RTV + FTC/TDF: FTC/TDF, darunavir (DRV), and RTV, orally, once daily.
  Emtricitabine/tenofovir disoproxil fumarate: A combination drug of two nucleoside reverse transcriptase inhibitors (NRTIs) Darunavir: A protease inhibitor (PI) Ritonavir: A protease inhibitor (PI)
Period: Overall Study
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Started | 605 | 603 | 601
Completed | 516 | 531 | 500
Not Completed | 89 | 72 | 101
Not completed — Death | 10 | 6 | 13
Not completed — Lost to Follow-up | 29 | 23 | 34
Not completed — Not able to get to clinic | 28 | 35 | 30
Not completed — Not willing to adhere to requirements | 12 | 2 | 16
Not completed — Withdraw consent prior study completion | 4 | 6 | 5
Not completed — Site Closure | 4 | 0 | 1
Not completed — Severe Debilitation | 2 | 0 | 1
Not completed — Complete Protocol: No follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat: All eligible participants were included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF | Total
Number analyzed (Participants) | 605 | 603 | 601 | 1809
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 2 | 6
  Between 18 and 65 years | 597 | 598 | 595 | 1790
  >=65 years | 6 | 3 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (11) | 37 (11) | 38 (11) | 37 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 148 | 143 | 435
  Male | 461 | 455 | 458 | 1374
Race/Ethnicity, Customized [Number; unit: participants] — Race/Ethnicity was collected prior to study entry
  participants
    White Non-Hispanic | 212 | 212 | 191 | 615
    Black Non-Hispanic | 252 | 254 | 251 | 757
    Hispanic (Regardless of Race) | 125 | 117 | 148 | 390
    Asian, Pacific Islander | 11 | 13 | 6 | 30
    American Indian, Alaskan Native | 2 | 2 | 2 | 6
    More than one race | 2 | 3 | 2 | 7
    Unknown/missing | 1 | 2 | 1 | 4
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] — HIV-1 RNA was calculated as the geometric mean of the two most recent HIV-1 RNA (log 10 copies/mL) obtained on or before study entry. In the event that these two values differed by more than 1log10 copy/mL, the outlying value (based on review of all HIV-1 RNA levels available prior to study entry by the study virologist) was excluded and baseline determined by the remaining sample. Note that screening HIV-1 RNA values were not sued in the calculation of baseline HIV-1 RNA levels.
  log10 copies/mL | 4.6 (0.7) | 4.6 (0.7) | 4.6 (0.7) | 4.6 (0.7)
CD4+ T-cell count [Mean (Standard Deviation); unit: cells/mm^3] — CD4+ T-cell counts were calculated as the mean of the two most recent values available on or before study entry.
  cells/mm^3 | 309 (189) | 306 (199) | 310 (189) | 308 (192)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Probability of First Virologic Failure by Week 96
Description: The Kaplan-Meier estimate of the cumulative probability of virologic failure by week 96.
  Time to virologic failure was defined as the first time from study entry to the first of two consecutive HIV-1 RNA >1000 copies/mL at or after week 16 and before week 24, or >200 copies/mL at or after week 24. Week 16 is defined to occur between 14 (98 days) and 18 weeks (126 days) after study entry, week 24 is defined to occur between 22 (154 days) and 26 (182 days) after study entry, and week 96 is defined to occur between 88 (616 days) and 104 (728 days) after study entry.
Time Frame: From study entry to week 96
Population: Intention to treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment.
Measure: Number (95% Confidence Interval); unit: cumulative probability per 100 persons
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
cumulative probability per 100 persons | 13 [10 to 16] | 10 [7 to 12] | 15 [12 to 18]
Statistical Analysis 1: Comparison: Arm A: ATV/RTV + FTC/TDF vs Arm B: RAL + FTC/TDF; Treatment comparison was made using the difference (arm A - arm B) in the stratified Kaplan-Meier estimate for the week 96 cumulative probability of virologic failure with 97.5% confidence interval; Test type: Non-Inferiority or Equivalence — Confidence interval estimation was stratified by HIV-1 RNA level at screening using Greenwood's variance with the inverse of this variance used for the stratum weights. The pre-specified confidence bounds for equivalence were +/-10 percentage points; Cumulative probability difference = 3.4, 97.5% CI 2-sided [-0.7 to 7.4]
Statistical Analysis 2: Comparison: Arm B: RAL + FTC/TDF vs Arm C: DRV/RTV + FTC/TDF; Treatment comparison was made using the difference (arm C - arm B) in the stratified Kaplan-Meier estimate for the week 96 cumulative probability of virologic failure with 97.5% confidence interval; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Cumulative probability difference = 5.6, 97.5% CI 2-sided [1.3 to 9.9]
Statistical Analysis 3: Comparison: Arm A: ATV/RTV + FTC/TDF vs Arm C: DRV/RTV + FTC/TDF; Treatment comparison was made using the difference (arm A - arm C) in the stratified Kaplan-Meier estimate for the week 96 cumulative probability of virologic failure with 97.5% confidence interval; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Cumulative probability difference = -2.2, 97.5% CI 2-sided [-6.7 to 2.3]

2. Primary Outcome: Cumulative Incidence of Discontinuation of the RAL or PI Component of Randomized Treatment for Toxicity by Week 96
Description: The cumulative incidence of discontinuation for toxicity by week 96 was estimated using competing risks with treatment discontinuation for other reasons considered as a competing event; participants completing the study on the RAL or PI component of their randomized regimen were considered censored at the earliest of the date of last patient contact and off study date.
Time Frame: From study entry to week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: cumulative events per 100 persons
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
cumulative events per 100 persons | 14 [12 to 17] | 1 [1 to 3] | 5 [3 to 7]
Statistical Analysis 1: Comparison: Arm A: ATV/RTV + FTC/TDF vs Arm B: RAL + FTC/TDF; Treatment comparison was made using the methods of Gray. Inference regarding comparisons of the treatment groups (arm A and arm B) with respect to equivalence was made based on the two-sided 97.5% confidence intervals of differences (arm A - arm B) in 96 week probability of tolerability failure with 97.5% confidence interval; Test type: Non-Inferiority or Equivalence — Although the study was not specifically powered to be able to detect equivalence, equivalence was declared if the 97.5% confidence interval difference in the cumulative probability of the tolerability endpoint by 96 weeks was entirely contained within +/-10 percentage points; Cumulative incidence difference = 12.8, 97.5% CI 2-sided [9.4 to 16.1]
Statistical Analysis 2: Comparison: Arm B: RAL + FTC/TDF vs Arm C: DRV/RTV + FTC/TDF; Treatment comparison was made using the methods of Gray. Inference regarding comparisons of the treatment groups (arm C and arm B) with respect to equivalence was made based on the two-sided 97.5% confidence intervals of differences (arm C - arm B) in 96 week probability of tolerability failure with 97.5% confidence interval; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Cumulative incidence difference = 3.6, 97.5% CI 2-sided [1.4 to 5.8]
Statistical Analysis 3: Comparison: Arm A: ATV/RTV + FTC/TDF vs Arm C: DRV/RTV + FTC/TDF; Treatment comparison was made using the methods of Gray. Inference regarding comparisons of the treatment groups (arm A and arm C) with respect to equivalence was made based on the two-sided 97.5% confidence intervals of differences (arm A - arm C) in 96 week probability of tolerability failure with 97.5% confidence interval; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Cumulative incidence difference = 9.2, 97.5% CI 2-sided [5.5 to 12.9]

3. Secondary Outcome: Cumulative Incidence of First Adverse Event by Week 96
Description: The cumulative incidence of first adverse event (with and without total bilirubin and creatine kinase and measured from study entry) by week 96 was estimated using methods for competing risks. Discontinuation of randomized treatment prior to an adverse event was considered a competing event.
  The time to the first of any post-entry Grade 2, 3, or 4 sign or symptom, or Grade 3 or 4 laboratory abnormality while on randomization. The protocol required reporting of signs and symptoms and laboratory values as follow: all signs and symptoms grade ≥2 post-entry to week 48, signs and symptoms grade >3 after week 48, and laboratory values grade >3 and all signs, symptoms, and laboratory values that led to a change in treatment, regardless of grade throughout out all post-entry follow-up.
Time Frame: From study entry to week 96
Population: As treated: Participants who had events occurring while on randomized treatment are included in this analysis: grade 2 events occurring in the after 48 weeks on study are excluded. Participants were analyzed per original assigned randomized treatment.
Measure: Number (95% Confidence Interval); unit: cumulative events per 100 persons
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 600 | 599 | 597
cumulative events per 100 persons | 81 [77 to 84] | 59 [55 to 63] | 65 [61 to 69]

4. Secondary Outcome: Cumulative Probability of Time to Loss of Virologic Response (TLOVR) by Week 96
Description: The Kaplan-Meier estimate of the cumulative probability of TROVR by week 96.
  A composite TLOVR endpoint defined in the CDER of the FDA document "Guidance for Industry - Antiretroviral Drugs Using Plasma HIV RNA Measurements - Clinical Consideration for Accelerated and Traditional Approval" (Appendix B, pages 20) http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm070968.pdf.
  If participants never achieved a confirmed HIV-1 RNA≤200 cp/mL (on two consecutive visits) prior to death, permanent discontinuation of randomized treatment, or time of last available HIV-1 RNA evaluation, TLOVR was equal to 0; otherwise, TLOVR was the earliest time of permanent discontinuation of randomized treatment prior to study close-out period, time to confirmed levels >200 cp/mL, or time to death. If TLOVR is immediately preceded by a single missing scheduled visit or multiple consecutive missing scheduled visits, TLOVR is replaced by the first such missing visit.
Time Frame: From study entry to week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: cumulative probability per 100 persons
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
cumulative probability per 100 persons | 31 [27 to 35] | 16 [14 to 19] | 24 [20 to 27]

5. Secondary Outcome: Presence of Mutations Associated With NRTI Resistance
Description: The number of participants with NRTI resistance determined by the Stanford resistance scoring algorithm (Version 6.3). All sequencing was performed regardless of status on randomized treatment at the time of virologic failure; no sequencing was performed on subjects not meeting virologic failure.
Time Frame: At the virologic failure at any time throughout the study (up to 213 weeks)
Population: Participants who met the criteria for virologic failure with successful sequencing at virologic failure
Measure: Number; unit: participants
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 75 | 65 | 99
participants | 8 | 7 | 3

6. Secondary Outcome: Presence of Mutations Associated With ATV/RTV or DRV/RTV Resistance
Description: The number of participants with ATV/RTV or DRV/RTV resistance determined by the Stanford resistance scoring algorithm (Version 6.3). All sequencing was performed regardless of status on randomized treatment at the time of virologic failure; no sequencing was performed on subjects not meeting virologic failure.
Time Frame: At the virologic failure at any time throughout the study (up to 213 weeks)
Population: Participants who met the criteria for virologic failure with successful sequencing at virologic failure
Measure: Number; unit: participants
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 75 | 65 | 99
participants | 0 | 0 | 0

7. Secondary Outcome: Presence of Mutations Associated With INI Resistance
Description: The number of participants with INI resistance determined by the Stanford resistance scoring algorithm (Version 6.3). All sequencing was performed regardless of status on randomized treatment at the time of virologic failure; no sequencing was performed on subjects not meeting virologic failure.
Time Frame: At the virologic failure at any time throughout the study (up to 213 weeks)
Population: Participants who met the criteria for virologic failure restricted to participants in the RAL group and random sample of participants in PI/RTV groups with successful sequencing at virologic failure.
Measure: Number; unit: participants
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 15 | 46 | 14
participants | 1 | 1 | 1

8. Secondary Outcome: CD4+ T-cell Count
Description: The absolute levels of CD4+ T-cell counts (cells/mm3)
Time Frame: At Weeks 24, 48, 96, and 144
Population: Intention to treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment. Missing data were assumed missing completely at random.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
cells/mm^3
  week 24 (nA=582, nB=574, nC=579) | 462 [443 to 480] | 460 [440 to 480] | 457 [438 to 476]
  week 48 (nA=564, nB=565, nC=559) | 524 [504 to 544] | 526 [504 to 549] | 509 [488 to 529]
  week 96 (nA=523, nB=541, nC=525) | 587 [565 to 609] | 596 [573 to 619] | 564 [541 to 586]
  week 144 (nA=395, nB=418, nC=394) | 622 [596 to 648] | 631 [602 to 660] | 596 [571 to 622]

9. Secondary Outcome: CD4+ T-cell Count Changes From Baseline
Description: Change was calculated as the CD4+ T-cell count at week (24, 48, 96, and 144) minus the baseline CD4+ T-cell count
Time Frame: Study entry to weeks 24, 48, 96, and 144
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
cells/mm^3
  week 24 (nA=582, nB=574, nC=579) | 157 [147 to 167] | 153 [142 to 163] | 147 [136 to 157]
  week 48 (nA=564, nB=565, nC=559) | 218 [206 to 231] | 218 [205 to 232] | 201 [187 to 214]
  week 96 (nA=523, nB=541, nC=525) | 284 [269 to 300] | 288 [272 to 304] | 256 [240 to 271]
  week 144 (nA=395, nB=418, nC=394) | 324 [305 to 343] | 325 [304 to 345] | 288 [269 to 307]

10. Secondary Outcome: Incidence of Death or AIDS Defining Events (CDC Category C)
Description: The incidence of death or AIDS defining events (CDC category C) was estimated as number of incident events over total person years of follow-up. Multiple new events for a single subject were counted toward events totals in estimation of event incidence; generalized estimating equations were used to estimation of robust standard errors for the incidence.
Time Frame: Study entry to off-study at any time throughout the study (up to 213 weeks), participant follow-up time was variable
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
events per 100 person-years | 1.55 [1.05 to 2.28] | 1.64 [1.12 to 2.40] | 2.14 [1.43 to 3.20]

11. Secondary Outcome: Incidence of Targeted Serious Non-AIDS Defining Events (Renal Failure, Liver Disease, Serious Metabolic Disorder, and CVD)
Description: The incidence of targeted serious non-AIDS defining events was estimated as number of incident events over total person years of follow-up. Multiple new events for a single subject were counted toward events totals in estimation of event incidence; generalized estimating equations were used to estimation of robust standard errors for the incidence.
Time Frame: Study entry to off-study at any time throughout the study (up to 213 weeks), participant follow-up time was variable
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: events per 100 person-years
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
events per 100 person-years | 2.38 [1.76 to 3.23] | 2.24 [1.51 to 3.32] | 2.69 [1.89 to 3.84]

12. Secondary Outcome: Change in Fasting Total Cholesterol Level From Baseline
Description: Only fasting results are included. Change was calculated as the fasting total cholesterol at week (48, 96, and 144) minus the baseline fasting total cholesterol.
Time Frame: Study entry to weeks 48, 96, and 144
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
mg/dL
  week 48 (nA=521, nB=542, nC=507) | 13 [10 to 16] | 1 [-2 to 3] | 15 [12 to 18]
  week 96 (nA=490, nB=505, nC=490) | 16 [13 to 19] | 3 [1 to 6] | 14 [11 to 17]
  week 144 (nA=364, nB=397, nC=363) | 20 [15 to 25] | 6 [2 to 9] | 19 [16 to 23]

13. Secondary Outcome: Change in Fasting HDL Cholesterol Level From Baseline
Description: Only fasting results are included. Change was calculated as the fasting HDL cholesterol at week (48, 96, and 144) minus the baseline fasting HDL cholesterol.
Time Frame: Study entry to weeks 48, 96, and 144
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
mg/dL
  week 48 (nA=522, nB=542, nC=506) | 6 [5 to 7] | 5 [4 to 6] | 5 [4 to 6]
  week 96 (nA=490, nB=505, nC=488) | 7 [5 to 8] | 6 [5 to 7] | 5 [4 to 6]
  week 144 (nA=364, nB=397, nC=363) | 8 [7 to 9] | 6 [5 to 7] | 7 [6 to 8]

14. Secondary Outcome: Change in Fasting Triglycerides Level From Baseline
Description: Only fasting results are included. Change was calculated as the fasting triglycerides at week (48, 96, and 144) minus the baseline fasting triglycerides.
Time Frame: Study entry to weeks 48, 96, and 144
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
mg/dL
  week 48 (nA=522, nB=542, nC=507) | 18 [11 to 24] | -9 [-16 to -3] | 16 [8 to 24]
  week 96 (nA=490, nB=505, nC=490) | 19 [12 to 27] | -9 [-16 to -1] | 16 [7 to 25]
  week 144 (nA=364, nB=397, nC=363) | 12 [4 to 19] | -4 [-13 to 4] | 20 [10 to 30]

15. Secondary Outcome: Change in Fasting Plasma Glucose Level From Baseline
Description: Only fasting results are included. Change was calculated as the fasting plasma glucose at week (48, 96, and 144) minus the baseline fasting plasma glucose.
Time Frame: Study entry to weeks 48, 96, and 144
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
mg/dL
  week 48 (nA=517, nB=535, nC=506) | 2.2 [0.7 to 3.8] | 1.3 [-0.3 to 2.8] | 2.1 [0.8 to 3.4]
  week 96 (nA=489, nB=499, nC=481) | 3.0 [1.4 to 4.6] | 0.9 [-0.6 to 2.5] | 2.5 [0.5 to 4.5]
  week 144 (nA=353, nB=392, nC=358) | 2.2 [-0.8 to 5.2] | 0.9 [-1.6 to 3.4] | 3.6 [1.1 to 6.0]

16. Secondary Outcome: Change in Framingham 10-year Risk of MI or Coronary Death From Baseline
Description: Only risk score estimated with fasting lipid results were included. Change was calculated as the Framingham 10-year risk of MI or coronary death at week (48, 96, and 144) minus the baseline Framingham 10-year risk of MI or coronary death. Framingham 10-year risk of MI or coronary death was calculated using Hear Coronary Heart Disease (10-year risk) found at https://www.framinghamheartstudy.org/risk-functions/coronary-heart-disease/hard-10-year-risk.php.
  Framingham 10-year risk of MI or coronary death was calculated according to age, laboratory values of total cholesterol and HDL cholesterol, smoking status, systolic blood pressure, and treatment for hypertension. The Framingham 10-year risk of MI or coronary death was calculated as: for males: <0 point (<1 percent risk) up to ≥17 points (≥30 percent risk); whereas for females: <9 points (<1 percent risk) up to ≥25 points (≥30 percent risk). Higher scores indicate high cardiovascular risk.
Time Frame: Study entry to weeks 48, 96, and 144
Population: Intention to treat: All participants with fasting lipids data were included, complete-case approach.
Measure: Mean (95% Confidence Interval); unit: percent risk
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
percent risk
  week 48 (nA=509, nB=537, nC=492) | 0.4 [0.2 to 0.6] | 0.0 [-0.2 to 0.1] | 0.4 [0.2 to 0.6]
  week 96 (nA=479, nB=493, nC=470) | 0.5 [0.3 to 0.7] | 0.2 [0.0 to 0.4] | 0.4 [0.2 to 0.6]
  week 144 (nA=347, nB=383, nC=349) | 0.6 [0.3 to 0.8] | 0.4 [0.2 to 0.7] | 0.9 [0.6 to 1.2]

17. Secondary Outcome: Change in Waist Circumference From Baseline
Description: Change was calculated as the waist circumference (based on mid-waist circumference) at week (48, 96, and 144) minus the baseline waist circumference.
Time Frame: Study entry to weeks 48, 96, and 144
Population: Intention to treat: All participants with waist circumference data were included, complete-case approach.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
cm
  week 48 (nA=555, nB=551, nC=547) | 2.3 [1.7 to 2.9] | 3.1 [2.5 to 3.7] | 2.1 [1.5 to 2.6]
  week 96 (nA=512, nB=526, nC=517) | 3.3 [2.6 to 4.0] | 4.0 [3.3 to 4.7] | 2.8 [2.2 to 3.5]
  week 144 (nA=425, nB=419, nC=409) | 3.6 [2.9 to 4.4] | 4.0 [3.2 to 4.8] | 3.4 [2.7 to 4.2]

18. Secondary Outcome: Change in Waist:Height Ratio From Baseline
Description: Change was calculated as the waist:height ratio at week (48, 96, and 144) minus the baseline waist:height ratio.
Time Frame: Study entry to weeks 48, 96, and 144
Population: Intention to treat: All participants with waist circumference data were included, complete-case approach.
Measure: Mean (95% Confidence Interval); unit: cm:cm
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
cm:cm
  week 48 (nA=555, nB=551, nC=547) | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.02] | 0.01 [0.01 to 0.02]
  week 96 (nA=512, nB=526, nC=517) | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.03] | 0.02 [0.01 to 0.02]
  week 144 (nA=425, nB=419, nC=409) | 0.02 [0.02 to 0.03] | 0.02 [0.02 to 0.03] | 0.02 [0.02 to 0.02]

19. Secondary Outcome: Self-reported Adherence
Description: Self-reported percentage of anti-HIV medications participant had taken during the last month at weeks 4, 24, 48, 96, and 144.
Time Frame: At Weeks 4, 24, 48, 96, and 144
Population: Intention to treat: All participants with fasting self-reported adherence data were included.
Measure: Mean (95% Confidence Interval); unit: percentage of prescribed medication
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Number analyzed (Participants) | 605 | 603 | 601
percentage of prescribed medication
  week 4 (nA=584, nB=590, nC=583) | 98 [98 to 99] | 97 [97 to 98] | 98 [98 to 99]
  week 24 (nA=570, nB=568, nC=562) | 97 [96 to 98] | 97 [96 to 97] | 96 [95 to 97]
  week 48 (nA=555, nB=547, nC=536) | 96 [95 to 97] | 97 [96 to 97] | 96 [95 to 97]
  week 96 (nA=508, nB=525, nC=507) | 96 [94 to 97] | 96 [95 to 97] | 96 [95 to 97]
  week 144 (nA=361, nB=376, nC=350) | 97 [96 to 98] | 97 [96 to 97] | 98 [97 to 98]

ADVERSE EVENTS:
Time Frame: From treatment dispensation until off-study at any time throughout the study (up to 213 weeks), participant follow-up time was variable
Description: The DAIDS Adverse Event (AE) Grading Table, Version 1.0, December 2004 (Clarification, August 2009) was used for grading of AEs. Expedited adverse event reporting followed "Manual for Expedited Reporting of Adverse Events to DAIDS" (DAIDS EAE Manual), dated May 6, 2004.
  MedDRA version 17.0
Arm/Group | Arm A: ATV/RTV + FTC/TDF | Arm B: RAL + FTC/TDF | Arm C: DRV/RTV + FTC/TDF
Serious Adverse Events (participants affected / at risk) | 139/605 | 126/603 | 125/601
Other Adverse Events (participants affected / at risk) | 565/605 | 516/603 | 532/601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: ATV/RTV + FTC/TDF (N=605) | Arm B: RAL + FTC/TDF (N=603) | Arm C: DRV/RTV + FTC/TDF (N=601)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Necrotising granulomatous lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0
Thyroid disorder (Endocrine disorders) | 0 | 1 | 0
Thyrotoxic crisis (Endocrine disorders) | 1 | 0 | 0
Eye disorder (Eye disorders) | 1 | 0 | 0
Necrotising retinitis (Eye disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1
Chest pain (General disorders) | 7 | 7 | 2
Cyst rupture (General disorders) | 0 | 0 | 1
Death (General disorders) | 3 | 1 | 2
Fatigue (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 4 | 3
Ulcer (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 0 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 1 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 4 | 1 | 3
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 2
Arthritis infective (Infections and infestations) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 2
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 6 | 5 | 5
Cryptococcosis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 0 | 1
Disseminated cytomegaloviral infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 2
Ear infection (Infections and infestations) | 1 | 0 | 0
Eye infection syphilitic (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 2
Hepatitis syphilitic (Infections and infestations) | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 2
Malaria (Infections and infestations) | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 1
Meningitis cryptococcal (Infections and infestations) | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 1 | 0
Mycobacterial infection (Infections and infestations) | 1 | 1 | 1
Neurosyphilis (Infections and infestations) | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis bacterial (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 8 | 6 | 8
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Proctitis herpes (Infections and infestations) | 0 | 1 | 0
Prostatic abscess (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 2 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Secondary syphilis (Infections and infestations) | 3 | 0 | 0
Sepsis (Infections and infestations) | 0 | 3 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 2
Viral myocarditis (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laryngeal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 3 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1
Chest X-ray abnormal (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 1 | 1
Laboratory test abnormal (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 2 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 2
Staphylococcus test positive (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Large cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 2
Complex partial seizures (Nervous system disorders) | 0 | 1 | 1
Complicated migraine (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1 | 1
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 3 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Wernicke's encephalopathy (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Catatonia (Psychiatric disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 6 | 4 | 4
Drug abuse (Psychiatric disorders) | 0 | 0 | 2
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 1
Homicidal ideation (Psychiatric disorders) | 1 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 0 | 2
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 2 | 0
Substance abuse (Psychiatric disorders) | 1 | 2 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 2 | 9
Suicide attempt (Psychiatric disorders) | 4 | 7 | 6
Nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 3 | 4
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alcohol detoxification (Surgical and medical procedures) | 0 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1 | 0 | 0
Cyst removal (Surgical and medical procedures) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Mastectomy (Surgical and medical procedures) | 0 | 0 | 1
Nephrectomy (Surgical and medical procedures) | 1 | 0 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 1 | 0 | 0
Spinal laminectomy (Surgical and medical procedures) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: ATV/RTV + FTC/TDF (N=605) | Arm B: RAL + FTC/TDF (N=603) | Arm C: DRV/RTV + FTC/TDF (N=601)
Ocular icterus (Eye disorders) | 40 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 35 | 23 | 32
Anogenital dysplasia (Gastrointestinal disorders) | 31 | 25 | 23
Diarrhoea (Gastrointestinal disorders) | 61 | 45 | 67
Nausea (Gastrointestinal disorders) | 61 | 43 | 59
Vomiting (Gastrointestinal disorders) | 42 | 29 | 40
Fatigue (General disorders) | 41 | 36 | 35
Pyrexia (General disorders) | 37 | 39 | 37
Bronchitis (Infections and infestations) | 28 | 33 | 28
Upper respiratory tract infection (Infections and infestations) | 36 | 28 | 29
Alanine aminotransferase increased (Investigations) | 68 | 59 | 46
Aspartate aminotransferase increased (Investigations) | 73 | 77 | 69
Blood bilirubin increased (Investigations) | 318 | 20 | 12
Blood cholesterol increased (Investigations) | 212 | 152 | 227
Blood creatinine increased (Investigations) | 105 | 73 | 98
Blood glucose decreased (Investigations) | 65 | 89 | 82
Blood glucose increased (Investigations) | 115 | 95 | 105
Blood phosphorus decreased (Investigations) | 70 | 67 | 70
Blood sodium decreased (Investigations) | 57 | 65 | 55
Low density lipoprotein increased (Investigations) | 184 | 139 | 183
Neutrophil count decreased (Investigations) | 74 | 85 | 74
Platelet count decreased (Investigations) | 25 | 32 | 24
White blood cell count decreased (Investigations) | 34 | 35 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 29 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 33 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 | 49 | 35
Headache (Nervous system disorders) | 45 | 48 | 46
Depression (Psychiatric disorders) | 47 | 60 | 53
Cough (Respiratory, thoracic and mediastinal disorders) | 54 | 53 | 46
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 32 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.